CLINICAL TRIAL: NCT04820127
Title: Personalized Management of Psycho-behavioral Symptoms in Alzheimer's Disease and Related Disorders: Impact on Health Resources Use
Brief Title: Personalized Management of Psycho-behavioral Symptoms in Alzheimer's Disease: Impact on Health Resources Use
Acronym: PERSON-AL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/19/0555
Record Dates: First submitted 2020-12-24; First posted 2021-03-29 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (usual care) (No Intervention): Patients in the control group will benefit from the usual care with a half-yearly visit by the specialist physician (geriatrician, neurologist or psychiatrist) according to AD French national management guidelines (HAS 2011 and HAS 2018).
- Intervention (personalized care program) (Experimental): Patients in the intervention group will benefit from personalized care preceded by a standardized assessment
  Interventions: Behavioral: personalized care preceded by a standardized assessment

INTERVENTIONS:
Behavioral: personalized care preceded by a standardized assessment — * personalized intervention plan (PIP) proposed to the patient/caregiver dyad to correct potentially reversible causes of psycho-behavioral symptoms. This PIP will be re-evaluated and adapted at each visit by the nurse in close collaboration with the GP;
  * PIP implementation will be based on a close follow-up during the 18 months follow-up coordinated by the nurse (3 memory consultation visits, 3 home visits (with the GP) and 6 phone calls). This follow up will be enhanced with the use of a web platform (allowing teleconsultation, tele-expertise and telemonitoring);
  * specific training on psycho-behavioral symptoms for caregivers at baseline and during follow-up will be performed. On line training on psycho-behavioral symptoms management for GP will be available;
  Arms: Intervention (personalized care program)

SUMMARY:
The present project propose to study the effectiveness of a personalized care management of psycho-behavioral symptoms based on an evidence-based standardized assessment to identify and understand the underlying causes of psycho-behavioral symptoms followed by a personalized intervention based on targeted and prioritized actions. This personalized intervention is proposed both to Alzheimer disease (AD) patients living at home with agitation-type psycho-behavioral symptoms, and also to their caregivers with the support and coordination of a nurse working in collaboration with the specialist physician and the General Practitioner (GP). News technologies are used to enhance the follow-up, based on telehealth, and caregiver training.

The project hypothesize that, for a vulnerable population at risk (AD patient with agitation and their caregivers) living at home, a personalized intervention, carried out and coordinated by a nurse in close collaboration with the specialist and GP, would reduce hospitalizations and have a positive effect on the disease evolution and caregiver distress. Also this personalized intervention could reduce the cost of care, in particular by reducing the costs associated with hospitalizations and informal help.

DETAILED DESCRIPTION:
PERSON-AL is a multicentric, interventional, open-label, randomized, parallel-group, stratified by centre, study comparing two arms: usual care versus intervention (personalized care preceded by a standardized assessment)

Principal Objective : To evaluate the impact of a personalized intervention for the management of agitation due to psycho-behavioral symptoms on the use of scheduled and unscheduled hospitalizations at 18 months in patients with AD and related disorders.

Secondary Objectives:

A- To evaluate the impact of a personalized intervention at 18 months on:

For the patient:

1. Unscheduled hospitalizations,
2. Severity of agitation symptoms,
3. The frequency and severity of emerging psycho-behavioral symptoms, other than agitation,
4. Prescription of psychotropic drugs,
5. Quality of life.

   For the caregiver:
6. Distress related to psycho-behavioral symptoms,
7. All causes hospitalizations,
8. Quality of life.

B- Evaluate the medico-economic impact of this personalized intervention, and in particular:

1. Its efficiency compared to usual management by means of cost-effectiveness and cost-utility analyses, from the community perspective and over a time horizon of 18 months,
2. The actual cost of patient's standardized assessment and personalized management
3. The use of care and associated costs for the caregiver and the efficiency of caregiver targeted intervention.

ELIGIBILITY:
Inclusion Criteria:

For the patient :

* Diagnosed with major neuro-cognitive disorders (DSM V) at all severity stages.
* Leaving at home
* Assisted by a caregiver, from patient's family or personal environment, assuming most of patient care (spending at least 6 hours per week with the patient)
* caregiver available to come with the patient to study visits as planned per protocol
* existing agitation since at least one month (according to International Psychogeriatric Association (IPA) criteria)
* agitation severity ≥ 2 , based on Clinician Global Impression of Severity (CGI-S) (at least mild severity)
* the patient, his/her family member/trusted person , or his /her legal responsible has provided written informed consent to participate in the study
* referring physician's oral approval obtained for patient participation in the study
* Affiliated to French Healthcare System

For the caregiver:

* Has provided his/her written informed consent to participate in the study
* Ability to understand and speak French properly, ability to complete the questionnaires and assess the patient.
* Affiliated to French Healthcare System

Exclusion Criteria:

For the patient:

* Agitation symptoms attributable either to other concomitant prescriptions, or to other psychiatric or evolving somatic diseases.
* Patient living in a residential care facility or having an institutionalization project within 6 months
* Patient with clinically significant or unstable disease that could affect he/her ability to come for the study visit or complete the evaluations planned as per protocol
* Concomitant participation to any other interventional research study
* Patient under legal protection.

For the caregiver:

* Caregiver under legal protection.
* Limited internet access or caregiver feeling unable to use it

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-10-14 (Estimated)

PRIMARY OUTCOMES:
patient's number of hospitalization at 18 months | From the inclusion until End of Study, 18 months
  number of all causes hospitalization, either scheduled or unscheduled, including emergency department visits

SECONDARY OUTCOMES:
patient's unscheduled hospitalization | From the inclusion until End of Study, 18 months
  all causes hospitalization, unscheduled, including emergency department visits

OTHER OUTCOMES:
Patient agitation symptoms severity | From the inclusion until End of Study, 18 months
  assessed by Neuropsychiatric Inventory Clinician (NPI-C) scale based on the International Psychogeriatrics Association (IPA) (NPI-C-IPA) and Cohen-Mansfield Agitation Inventory (CMAI).
severity and frequency of others emergent psycho-behavioral symptoms | From the inclusion until End of Study, 18 months
  assessed by the NPI scale
  Frequency (0-4) Severity (0-3): Caregiver Distress (0-5):
Number of psychotropic drug prescription for the patient | From the inclusion until End of Study, 18 months
  prescription checked at each visit
patient's quality of life | From the inclusion until End of Study, 18 months
  assessed by the Euro Quality of life (EQ-5D-5L) scale
Patient's psycho-behavioral symptoms distress on the caregiver | From the inclusion until End of Study, 18 months
  "distress" score of the Neuropsychiatric Inventory-Clinician rating scale-IPA scale
  Frequency (0-4) Severity (0-3): Caregiver Distress (0-5):
caregiver's hospitalizations | From the inclusion until End of Study, 18 months
  all causes of hospitalization, either scheduled or unscheduled, including emergency department visits
caregiver's quality of life | From the inclusion until End of Study, 18 months
  assessed by the Euro Qol (EQ-5D-5L) scale
Cost/efficiency ratio and cost /utility differential from the community perspective | From the inclusion until End of Study, 18 months
  Cost/efficiency ratio and cost /utility differential from the community perspective
Comparison between Standardized evaluation and personalized care program real cost | From the inclusion until End of Study, 18 months
  micro-costing approach of health costs
quantity and cost health system resources used by the patient | From the inclusion until End of Study, 18 months
  health system resources used by the patient quantity and cost in comparison with efficiency and cost from the community perspective.
efficiency and cost from the community perspective. | From the inclusion until End of Study, 18 months
  health system resources used by the patient quantity and cost in comparison with efficiency and cost from the community perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Maria SOTO, MD, Principal Investigator — University Hospital Toulouse - Gerontopole
Locations (16):
- France (16):
  - CH d'Albi, Albi
  - CH de Cahors, Cahors
  - Carcassonne Hospital, Carcassonne
  - CHI Castres Mazamet, Castres
  - CH Lannemezan, Lannemezan
  - CH Lavaur, Lavaur
  - Limoges university hospital, Limoges
  - Lyon University Hospital, Lyon
  - CH Montauban, Montauban
  - Narbonne Hospital, Narbonne
  - Perpignan Hospital, Perpignan
  - CHI Val d'Ariège, Saint-Girons
  - Toulouse University Hospital (CHU de Toulouse), Toulouse
  - University Hospital Toulouse - Neurology department, Toulouse
  - CH de Bigorre, Vic-en-Bigorre
  - HNO-Franche-sur-Soâne, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No